CLINICAL TRIAL: NCT04842448
Title: Hyperbaric Oxygen for Treatment of Long COVID Syndrome; A Randomized, Placebo-Controlled, Double-Blind, Phase II Clinical Trial
Brief Title: Safety and Efficacy of Hyperbaric Oxygen Therapy for Long COVID Syndrome
Acronym: HOT-LoCO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other); Karolinska Trial Alliance (Industry); EDC Scandinavia AB (Unknown); Swedish Heart Lung Foundation (Other); Region Stockholm (Other Government); The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Anders Kjellberg, MD, ICU Consultant, head of hyperbaric medicine, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HOT-LoCO; 2021-000764-30 (EudraCT Number); K 2021-1592 (Other: Karolinska University Hospital); 4-621/2021 (Other: Karolinska Institutet); 2022-00834 (Other Grant/Funding Number: Swedish Research Council- Vetenskapsrådet); RS 2022-0674 (Other Grant/Funding Number: Region Stockholm)
Record Dates: First submitted 2021-04-09; First posted 2021-04-13 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: COVID-19; Post COVID-19 Condition; Post COVID-19 Condition, Unspecified; Post COVID Condition; Post-COVID Syndrome; Post-Acute COVID-19 Syndrome
Keywords: Long COVID; Post COVID Syndrome; COVID-19; Hyperbaric Oxygen; HBOT; Health Related Quality of Life; Endothelial dysfunction
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind, phase II
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized to either active treatment or sham treatment. Assessors will be blinded to treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperbaric oxygen treatment (Experimental): HBO2 240 kPa, 90 min, maximum 10 treatments
  Interventions: Drug: Hyperbaric oxygen
- Sham treatment (Placebo Comparator): Air 134-120 kPa, 90 min, maximum 10 treatments
  Interventions: Procedure: Sham treatment

INTERVENTIONS:
Drug: Hyperbaric oxygen — Hyperbaric oxygen 240 kPa for 90 minutes (with 10 min compression time, 2 air bakes and 10 minutes decompression time).
  Other Names: HBO; HBO2; HBOT
  Arms: Hyperbaric oxygen treatment
Procedure: Sham treatment — Sham treatment 134-120 kPa Air (with 5 min compression time, and 5 min decompression to 120 kPa, two air brakes will be reported to the subjects)
  Other Names: Placebo
  Arms: Sham treatment

SUMMARY:
Long COVID Syndrome (Long COVID), Post Acute COVID-19 Syndrome (PACS) or Post COVID-19 Syndrome (PCS) is defined as 'signs and symptoms that develop during or following an infection consistent with COVID-19, continue for more than 12 weeks and are not explained by an alternative diagnosis'. 1 in 10 infected individuals may suffer persistent symptoms, and we are facing an emerging problem that will severely affect individuals, health care systems and society for years to come.

We explore hyperbaric oxygen administered in a randomized placebo-controlled clinical trial as a potential treatment for patients suffering from Long COVID.

The overall hypothesis to be evaluated is that hyperbaric oxygen (HBO2) alleviates symptoms associated with Long COVID.

DETAILED DESCRIPTION:
Phase II Clinical Trial

Prospective randomized, placebo-controlled, double blind, phase II, clinical trial, estimated enrolment: 80 subjects Parallel groups Intervention: HBO2: 240 kPa for 90 min, maximum 10 treatments within 6 weeks from randomization

Control: Placebo treatment with 'sham' air breathing at a moderately higher pressure (134 kPa) to simulate hyperbaric chamber treatment, maximum 10 treatments within 6 weeks from randomization

The population will comprise of previously healthy patients (American Society of Anaesthesiologists (ASA) class 1-2 diagnosed with Long COVID (U09.9) by a multidisciplinary team. All patients are assessed with a battery of questionnaires, physical tests, laboratory tests and radiology. After their first assessment, individuals may have further organ specific work up for diagnosis, such as diagnosis of Postural Orthostatic Tachycardia Syndrome (POTS).

Once the patient has been diagnosed with Long COVID, they will be informed and asked to participate in the trial. No study specific procedures will take place before an informed consent form (ICF) has been signed. The patients will be included once they fulfil the inclusion criteria and exhibit none of the exclusion criteria. Some study specific procedures will be performed before inclusion. Eligible subjects will be randomized within two weeks of the planned first treatment. Subjects will be randomized in a 1:1 allocation to HBO2 or placebo (sham treatment). Scheduling of the HBOT will depend on available resources but the first treatment should be given within two weeks after randomization, and a maximum ten treatments should be given within 6 weeks from randomization.

Clinical equipoise: The rationale for 1:1 randomization is that this is a new disease and that it will maximise the statistical power to detect a statistically significant efficacy between treatment groups.

Main efficacy and safety endpoints will be evaluated at three months but the trial will continue for one year after inclusion or until withdrawal. There will also be a four year post-trial follow up of health-economy.

The trial will be conducted in compliance with Good Clinical Practice (GCP), the Declaration of Helsinki and national regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-60 years
2. Healthy or mild systemic disease (ASA 1-2) prior to COVID-19
3. Symptoms consistent with Long COVID for at least 12 weeks
4. Diagnosed with Long COVID, PACS, PCS (ICD-10 U09.9)
5. Working or studying prior to COVID-19
6. Documented informed consent according to GCP and national regulations

Exclusion Criteria:

1. Known pregnancy or positive pregnancy test in women of childbearing age
2. ASA 3 or more from other cause than Long COVID
3. Score above 70 in RAND-36 Role Limitation Physical Health (RP) or Physical Functioning (PF)
4. Diabetes
5. Diagnosed with hypertension prior to COVID-19
6. Contraindication for hyperbaric oxygen treatment according to local guidelines
7. Participation or recent participation in a clinical trial with an investigational product
8. Mental inability, reluctance or language difficulties that result in difficulty understanding the meaning of study participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
RAND 36 change | Baseline and 13 weeks
  Mean change from baseline to 13 weeks in RAND 36 domains role limitations due to physical health (RP) and physical functioning (PF).
  RAND 36 is a self-reporting questionnaire that contains 36 items that measure eight concepts of health in general terms, at present and past four weeks. Numeric values from the survey are coded so that all items are scored from 0 (lowest score) to 100 (highest possible score). Scores then represent the percentage of total possible score achieved. Items in the same scale are averaged together to create the eight scale scores. Items that are left blank (missing data) are not taken into account when calculating the scale scores. Hence, scale scores represent the average for all items in the scale that the respondent answered.

SECONDARY OUTCOMES:
Endothelial dysfunction | Baseline and 13 weeks
  Mean change from baseline to 13 weeks in Reactive Hyperemia Index (RHI)
6-min walk test | Baseline and 13 weeks
  Mean change from baseline to 13 weeks in the 6-min walk test
30/60 min chair stand | Baseline and 13 weeks
  Mean change from baseline to 13 weeks in the 30/60 sec chair stand
EQ-5D | Baseline and 13 weeks
  Mean change from baseline to 13 weeks in EQ-5D.
  EuroQol-5 Dimensions questionnaire is a widely used self-reporting questionnaire that measure 5 dimensions of health TODAY at three or five levels (EQ-5D-3L or EQ-5D-5L) of severity; no problems, some/moderate problems and extreme problems/unable.The health dimensions are mobility, self-care, usual activities, pain/discomfort, anxiety/depression and a visual analogue scale (VAS) 0-100 which it used as a quantitative measure of overall health status. EQ-5D is the most widely used questionnaire for health-economic evaluation.
RAND 36 normalization | Baseline and 13 weeks
  Proportion of subjects with a normalisation of levels in RAND-36 domains role limitations due to physical health and physical functioning respectively, at 13 weeks.

OTHER OUTCOMES:
Adverse Events (AE) | Baseline and 13 weeks
  Number of AEs at 13 weeks.
Compliance | Baseline and 13 weeks
  Number of subjects, proportion of subjects that have completed planned treatments and number of treatments after 6 weeks.
RAND 36 longitudinal | Baseline, 13 weeks, 26 weeks and 52 weeks
  Mean change in other RAND 36 domains at 13, 26 and 52 weeks compared to baseline.
EQ-5D Health economy | Baseline, 6 weeks, 26 weeks and 52 weeks
  Mean change in EQ-5D at 6, 26 and 52 weeks compared to baseline.
Physical activity | Baseline, 6 weeks, 13 weeks and 26 weeks
  Mean change in physical activity using an activity meter at 6, 13 and 26 weeks compared to baseline
Heart Rate Variability (HRV) | Baseline, 6 weeks, 13 weeks and 26 weeks
  Mean change in HRV using an activity meter at 6, 13 and 26 weeks compared to baseline
Restorative sleep | Baseline, 6 weeks, 13 weeks and 26 weeks
  Mean change in sleeping pattern using an activity meter at 6, 13 and 26 weeks compared to baseline.
Hypoxia response | Baseline, 6 weeks, 13 weeks and 26 weeks
  Mean change from baseline in hypoxia pathways in PBMCs evaluated by RNA sequencing, at 6, 13 and 26 weeks.
Inflammatory response | Baseline, 6 weeks, 13 weeks and 26 weeks
  Mean change from baseline in inflammatory pathways in PBMCs evaluated by RNA sequencing, at 6, 13 and 26 weeks
Redox status | Baseline, 6 weeks and 13 weeks
  Mean change from baseline of reactive oxygen species in red blood cells measured by Electron paramagnetic resonance spectroscopy (EPR) at 6 and 13 weeks.
Long term follow-up RAND-36 | Baseline, 26 weeks and 52 weeks
  Long-term follow up of change in HRQoL with self-reported questionnaire RAND-36
Health-economic evaluation | Baseline, 13 weks, 26 weeks and 52 weeks
  Economical cost/benefit evaluation using EQ-5D as variable
microRNA | Baseline, 6 weeks and 13 weeks
  Mean change from baseline of microRNA in plasma, at 6 and 13 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Kjellberg, MD, PhD, Principal Investigator — Karolinska University Hospital (and Karolinska Insitutet); Judith Bruchfeld, MD, PhD, Study Chair — Karolinska University Hospital (and Karolinska Insitutet); Malin Nygren-Bonnier, PhD, Study Chair — Karolinska University Hospital (and Karolinska Insitutet); Michael Runold, MD, PhD, Study Chair — Karolinska University Hospital (and Karolinska Insitutet); Marcus Ståhlberg, MD, PhD, Study Chair — Karolinska University Hospital (and Karolinska Insitutet); Peter Lindholm, MD, PhD, Study Chair — Karolinska Insitutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The full study protocol, statistical plan and consent form will be publicly available. Data will be available on patient level; data will be pseudonymized, the full dataset and statistical code will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after study completion and for 36 months
Access Criteria: A full description of the intended use of the data must be sent to the corresponding author for review and approval. Participant consent for data sharing is conditioned and new ethics approval may be required.

REFERENCES:
- [Background] Venkatesan P. NICE guideline on long COVID. Lancet Respir Med. 2021 Feb;9(2):129. doi: 10.1016/S2213-2600(21)00031-X. Epub 2021 Jan 13. No abstract available. PMID 33453162
- [Background] Dani M, Dirksen A, Taraborrelli P, Torocastro M, Panagopoulos D, Sutton R, Lim PB. Autonomic dysfunction in 'long COVID': rationale, physiology and management strategies. Clin Med (Lond). 2021 Jan;21(1):e63-e67. doi: 10.7861/clinmed.2020-0896. Epub 2020 Nov 26. PMID 33243837
- [Background] Kjellberg A, De Maio A, Lindholm P. Can hyperbaric oxygen safely serve as an anti-inflammatory treatment for COVID-19? Med Hypotheses. 2020 Nov;144:110224. doi: 10.1016/j.mehy.2020.110224. Epub 2020 Aug 30. PMID 33254531
- [Background] Kjellberg A, Abdel-Halim L, Hassler A, El Gharbi S, Al-Ezerjawi S, Bostrom E, Sundberg CJ, Pernow J, Medson K, Kowalski JH, Rodriguez-Wallberg KA, Zheng X, Catrina S, Runold M, Stahlberg M, Bruchfeld J, Nygren-Bonnier M, Lindholm P. Hyperbaric oxygen for treatment of long COVID-19 syndrome (HOT-LoCO): protocol for a randomised, placebo-controlled, double-blind, phase II clinical trial. BMJ Open. 2022 Nov 2;12(11):e061870. doi: 10.1136/bmjopen-2022-061870. PMID 36323462
- [Derived] Kjellberg A, Hassler A, Bostrom E, El Gharbi S, Al-Ezerjawi S, Schening A, Fischer K, Kowalski JH, Rodriguez-Wallberg KA, Bruchfeld J, Stahlberg M, Nygren-Bonnier M, Runold M, Lindholm P. Ten sessions of hyperbaric oxygen versus sham treatment in patients with long covid (HOT-LoCO): a randomised, placebo-controlled, double-blind, phase II trial. BMJ Open. 2025 Apr 14;15(4):e094386. doi: 10.1136/bmjopen-2024-094386. PMID 40228859
- [Derived] Kjellberg A, Hassler A, Bostrom E, El Gharbi S, Al-Ezerjawi S, Kowalski J, Rodriguez-Wallberg KA, Bruchfeld J, Stahlberg M, Nygren-Bonnier M, Runold M, Lindholm P. Hyperbaric oxygen therapy for long COVID (HOT-LoCO), an interim safety report from a randomised controlled trial. BMC Infect Dis. 2023 Jan 20;23(1):33. doi: 10.1186/s12879-023-08002-8. PMID 36670365
- See also: Research group Hyperbaric Medicine at Karolinska Institutet — https://ki.se/en/fyfa/hyperbaric-medicine